CLINICAL TRIAL: NCT03685955
Title: The Effect of Amniotic Membranes on Complex Genitourinary Reconstruction Outcomes in Pediatric and Adult Populations
Brief Title: Efficacy of Amniotic Membranes in Complex Genitourinary Reconstruction
Status: Withdrawn | Type: Observational
Why Stopped: Lack of supporting staff
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00168089
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hypospadias; Hypospadias and Epispadias and Other Penile Anomalies; Fistula; Fistula, Urinary; Bladder Exstrophy and Epispadias Complex; Bladder and Bladder Neck Disorders (Excluding Calculi)
MeSH Terms: conditions — Hypospadias; Epispadias; Fistula; Urinary Fistula; Bladder Exstrophy and Epispadias Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Genitourinary Reconstruction with Amniotic Membranes: Patients who undergo genitourinary reconstruction with amniotic membranes
  Interventions: Biological: Amniotic membranes

INTERVENTIONS:
Biological: Amniotic membranes — Amniotic membranes will be employed during participant's genitourinary reconstruction

SUMMARY:
Urinary fistulas are unfortunately one of the most common post operative complications in hypospadias repairs and bladder neck transections on pediatric and adult populations, an estimated 20%, resulting in multiple repeat operations with prolonged hospitalization. The negative sequelae of these fistulas have significant financial and psychosocial impact and the aim of this study is to evaluate if the fresh frozen preserved amniotic membrane tissue studied, which have live cells and intact naturally occurring growth hormones and peptides that augment healing that have been shown in early studies to be effective facilitating previous failed fistula repairs and leg ulcer healing, respectively, will help reduce the incidence of urinary fistulas in subject populations.

DETAILED DESCRIPTION:
Urinary fistulas in the pediatric and adult populations present significant surgical and economical challenges. These include urethrocutaneous and vesicocutaneous fistulas, which are unfortunately common in the investigators' patients with hypospadias and bladder exstrophy, respectively. Urethrocutaneous fistula is the most common complication following surgical repair of hypospadias with an incidence of 4-25%. This high complication rate is especially problematic as these fistulas once formed often recur requiring multiple surgical repairs resulting in potentially harmful physical and psychologic consequences on young patients. Vesicocutaneous fistulas develop in bladder exstrophy patients at a estimated rate of 20% following surgery aimed at making these patients continent by transecting the bladder neck and creating a catheterizable channel. Small, simple fistulas can be repaired primarily, however larger, multiple or recurrent fistulas must be closed in layers. Layered closures have been found to have higher success rates have been demonstrated with using additional tissue layers refistulization rate including local and distant tissue grafts, which add time and morbidity to surgical repairs.

Amniotic membranes have been shown to increase healing in chronic wounds such as a chronic venous stasis and diabetic ulcers and have been used in fistula repairs. Grafix and Stravix are frozen preserved placental membranes and Wharton's Jelly, respectively, that have high quantities of viable mesenchymal stem cells (MSCs), which add in tissue healing. The investigators believe these membranes can be used as a structural layer in fistula repairs, hypospadias repairs, and bladder neck closures to treat existing fistulas and prevent fistula formation in the primary repair setting.

1. This is a prospective study examining patients with hypospadias will be considered for repair with the use of amniotic membranes. The repair of fistula with graft tissue is standard of care.
2. Eligible patients will be identified in a clinic visit with one of the co-investigators.

   a. The patient will be consented and undergo a repair using amniotic membranes within the fistula site or primary repair at the discretion of the operating surgeon. Using different repair techniques is standard of care, however, the use of frozen preserved placental membranes is the study material. The size of the product will be determined by the surgical need at the time of repair.
3. The patient will be discharged be provided with routine postoperative care and seen in approximately 2 weeks per standard of are.
4. If the participant fails repair of participant's fistula, participant will not be offered a repeat repair with the amniotic membranes. Other forms of surgery may be offered, however.

ELIGIBILITY:
Inclusion Criteria:

* 6mo - 99 years old
* Undergoing surgical procedure with risk of or known urinary fistula

Exclusion Criteria:

* Failed prior repair with amniotic membranes
* Sensitivity to cryopreservation fluids or disinfecting solutions.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult populations with complex genitourinary reconstructive needs including pediatric hypospadias repair, bladder exstrophy, neurogenic bladder, urinary fistulas, urethral stricture disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Failure rate of complex genitourinary reconstruction after incorporation of placental membranes into repair. | 2 years
  We will evaluate patients with complex genitourinary wounds who have undergone surgical repair using preserved placental membranes, Grafix or Stravix. They will be evaluated in the standard post operative fashion to evaluate for failure of surgical repair of complex genitourinary reconstruction which will be defined by stricture recurrence, wound dehiscence, or recurrence of fistula.

CONTACTS AND LOCATIONS:
Overall Officials: Heather DiCarlo, MD, Principal Investigator — The Johns Hopkins School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frykberg RG, Gibbons GW, Walters JL, Wukich DK, Milstein FC. A prospective, multicentre, open-label, single-arm clinical trial for treatment of chronic complex diabetic foot wounds with exposed tendon and/or bone: positive clinical outcomes of viable cryopreserved human placental membrane. Int Wound J. 2017 Jun;14(3):569-577. doi: 10.1111/iwj.12649. Epub 2016 Aug 3. PMID 27489115
- [Background] Suzuki K, Michael G, Tamire Y. Viable intact cryopreserved human placental membrane for a non-surgical approach to closure in complex wounds. J Wound Care. 2016 Oct 1;25(Sup10):S25-S31. doi: 10.12968/jowc.2016.25.Sup10.S25. PMID 27681807
- [Background] Duan-Arnold Y, Gyurdieva A, Johnson A, Uveges TE, Jacobstein DA, Danilkovitch A. Retention of Endogenous Viable Cells Enhances the Anti-Inflammatory Activity of Cryopreserved Amnion. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):523-533. doi: 10.1089/wound.2015.0636. PMID 26401419
- [Background] Cooke M, Tan EK, Mandrycky C, He H, O'Connell J, Tseng SC. Comparison of cryopreserved amniotic membrane and umbilical cord tissue with dehydrated amniotic membrane/chorion tissue. J Wound Care. 2014 Oct;23(10):465-74, 476. doi: 10.12968/jowc.2014.23.10.465. PMID 25296347
- [Background] Batsali AK, Kastrinaki MC, Papadaki HA, Pontikoglou C. Mesenchymal stem cells derived from Wharton's Jelly of the umbilical cord: biological properties and emerging clinical applications. Curr Stem Cell Res Ther. 2013 Mar;8(2):144-55. doi: 10.2174/1574888x11308020005. PMID 23279098
- [Background] Johnson EL, Tassis EK, Michael GM, Whittinghill SG. Viable placental allograft as a biological dressing in the clinical management of full-thickness thermal occupational burns: Two case reports. Medicine (Baltimore). 2017 Dec;96(49):e9045. doi: 10.1097/MD.0000000000009045. PMID 29245303
- [Result] Lavery LA, Fulmer J, Shebetka KA, Regulski M, Vayser D, Fried D, Kashefsky H, Owings TM, Nadarajah J; Grafix Diabetic Foot Ulcer Study Group. The efficacy and safety of Grafix((R)) for the treatment of chronic diabetic foot ulcers: results of a multi-centre, controlled, randomised, blinded, clinical trial. Int Wound J. 2014 Oct;11(5):554-60. doi: 10.1111/iwj.12329. Epub 2014 Jul 21. PMID 25048468